CLINICAL TRIAL: NCT03741426
Title: WIndow of Opportunity Clinical Trials Platform for Evaluation of Novel Treatments Strategies in REnal Cell Cancer
Brief Title: WIRE - Novel Treatments in Renal Cell Cancer
Acronym: WIRE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: University of Cambridge (Other); AstraZeneca (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Prof. Grant D. Stewart, MBChB, BSc., FRCSEd (Urol), PhD, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: WIRE
Record Dates: First submitted 2018-10-31; First posted 2018-11-14 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Renal Cell Cancer
Keywords: Olaparib; Cediranib; Durvalumab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — olaparib; cediranib; durvalumab

STUDY DESIGN:
Intervention Model Description: Bayesian Adaptive
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1- Cediranib (Experimental): Cediranib tablet oral 20mg once daily for a minimum of 2 weeks up until 36 hours before nephrectomy.
  Interventions: Drug: Cediranib
- Arm 2- Olaparib (Experimental): Olaparib tablet oral 300mg twice daily for a minimum of 2 weeks up until the morning of nephrectomy.
  Interventions: Drug: Olaparib
- Arm 3- Olaparib and Cediranib (Active Comparator): Olaparib tablet oral 300mg twice daily for a minimum of 2 weeks up until the morning of nephrectomy AND Cediranib tablet oral 20mg once daily for a minimum of 2 weeks up until 36 hours before nephrectomy.
  Interventions: Drug: Olaparib; Drug: Cediranib
- Arm 4- Durvalumab (Experimental): Durvalumab 1500mg intravenous infusion once, a maximum of 4 weeks prior to nephrectomy.
  Interventions: Drug: Durvalumab
- Arm 5- Olaparib and Durvalumab (Active Comparator): Olaparib tablet oral 300mg twice daily for a minimum of 2 weeks up until the morning of nephrectomy. Durvalumab 1500mg intravenous infusion once, a maximum of 4 weeks prior to nephrectomy.
  Interventions: Drug: Olaparib; Drug: Durvalumab

INTERVENTIONS:
Drug: Olaparib — Olaparib 300mg twice daily, oral medication administered for at least 2 weeks and up until the morning of nephrectomy. Arms 2, 3 and 5
  Other Names: AZD2281; KU-0059436; LYNPARZA
  Arms: Arm 2- Olaparib; Arm 3- Olaparib and Cediranib; Arm 5- Olaparib and Durvalumab
Drug: Cediranib — Cediranib 20mg once daily, oral medication administered for at least 2 weeks until 36 hours prior to nephrectomy. Arms 1 and 3
  Other Names: AZD2171
  Arms: Arm 1- Cediranib; Arm 3- Olaparib and Cediranib
Drug: Durvalumab — Durvalumab 1500mg intravenous infusion administered once, no greater than 4 weeks prior to nephrectomy
  Other Names: MEDI4736
  Arms: Arm 4- Durvalumab; Arm 5- Olaparib and Durvalumab

SUMMARY:
Evaluation of proof of mechanism with relation to ktrans and/or CD8 count when 3 different IMPs are given as monotherapy or as combination therapy. These would be administered in the "window of opportunity", prior to nephrectomy in surgically resectable renal cell cancer

DETAILED DESCRIPTION:
A Phase 2, multi-arm, multicentre, non-randomised, proof-of-mechanism (single and combination IMPs) trial using a Bayesian adaptive design.

A multi-centre trial. 2 centres initially planned - this may be reduced or increased in order to recruit the required number of participants.

Up to sixty (60) patients with surgically resectable renal cell cancer (Stage M0/M1). Up to twelve (12) participants will be registered for each of the single treatment arms and up to twenty (20) participants for the combination treatment arm(s) as per the Bayesian adaptive design.

The trial duration consists of a 28 day screening period, a minimum of 2 weeks oral IMP (Olaparib and/or Cediranib) treatment or a single dose of durvalumab alone or in combination in the window-of-opportunity period prior to surgery (nephrectomy or partial nephrectomy) performed as standard of care.

Participants will continue oral IMP treatment up until surgery (stopping when indicated for surgical safety reasons). As such treatment duration will be variable and an optional 21 day telephone assessment will take place for patients who remain on IMP. Patients will then be reviewed in the surgical follow-up clinic at 6 weeks and 3 months post-surgery as standard of care.

For patients on monotherapy or combination Olaparib and Cediranib IMP, response will be measured using DCE-MRI (Ktrans), defining reduced tumour capillary permeability.

For patients on monotherapy Durvalumab, or combination Olaparib and Durvalumab, response will be measured using CD8 positive T cells.

Additional safety outcomes will be assessed, along with the tumour response and various biological measures that would indicate drug mechanistic response.

ELIGIBILITY:
Inclusion Criteria:

Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Aged ≥18 years and over. Predicted life expectancy ≥ 3 months. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1. Have biopsy proven clear cell RCC. Have a surgically resectable tumour as determined by the treating Urologist Have any T or N status, M0. Have any T or N status, M1 (but if M1, the subject must be deemed suitable for cytoreductive nephrectomy at time of enrolment).

No prior exposure to PARP inhibitors (including but not limited to olaparib), tyrosine kinase inhibitors (including but not limited to cediranib, sunitinib, pazopanib, axitinib or cabozantinib), immunotherapy or immune checkpoint inhibitors (including but not limited to other anti-CTLA-4, anti-PD-1, or anti-PD-L1 antibodies), nor prior treatment with an mammalian target of rapamycin (mTOR) inhibitor (including, but not limited to everolimus, temsirolimus, or sirolimus). Prior cytokine therapy (eg, IL-2, IFN-α) or treatment with cytotoxics is allowed.

At least 1 measurable lesion according to RECIST Version 1.1 at screening that can be accurately assessed at baseline by CT or MRI and is suitable for repeated assessment. A previously irradiated lesion cannot be considered a target lesion. Radiographic disease assessment can be performed up to 28 days prior to the first dose of trial treatment. It is acceptable for the measurable lesion to be planned for removal at surgery.

Have adequate organ and marrow function, as defined below (measured within 28 days of first dose of trial medication):

Haemoglobin ≥ 100 g/L Platelet count ≥ 135 x 109/L Neutrophil count ≥ 1.8 x 109/L Peripheral blood smear with no features of myelodysplastic syndrome or acute myeloid leukemia.

Serum creatinine ≤1.5x the institutional ULN concurrent with creatinine clearance ≥51mL/min (calculated by Cockcroft and Gault equation)

Adequate hepatic function:

Alanine Aminotransferase (ALT) ≤2.5x the institutional upper limit of normal (ULN) unless liver metastases are present, in which case it must be ≤5x the institutional ULN, AND Total bilirubin ≤1.5x the institutional ULN unless in the presence of Gilbert's syndrome (persistent or recurrent hyperbilirubinaemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology), AND

Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy) Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

For women of childbearing potential a negative urine or serum pregnancy test must be performed within 28 days of study treatment and confirmed prior to treatment on day 1.

Patient is willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

Patients with brain metastases. A scan to confirm the absence of brain metastases is not required.

Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.

History of leptomeningeal carcinomatosis. Body weight <30kg Contraindication to cediranib, olaparib, durvalumab or chimeric or humanized antibodies or fusion proteins.

Specifically patients with hereditary galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption should not enter the study.

History of hypersensitivity to active or inactive excipients of cediranib, olaparib or durvalumab.

Other invasive malignancy within the last 2 years. Patients with previous history of malignancies with a negligible risk of metastasis or death and treated with expected curative intent are eligible at discretion of clinical team, for example:

Carcinoma in situ of the cervix. Basal or squamous cell skin cancer. Localized low to intermediate risk prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse; or prostate cancer (Stage T1/T2a, Gleason ≤ 6 and PSA < 10 ng/mL) undergoing active surveillance and treatment naïve.

Major surgery within 4 weeks prior to first dose of study drug (excluding placement of vascular access).

Patients must have recovered from side effects of any major surgery. Minor surgery (not including the diagnostic biopsy) within 2 weeks prior to first dose of trial treatment.

Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

Concurrent enrollment in another clinical trial unless it is an observational (non-interventional) or translational clinical study, or during the follow-up period of an interventional clinical study.

Receipt of the last dose of anticancer therapy or radiotherapy chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolisation, monoclonal antibodies) ≤28 days prior to the first dose of study drug (If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca/MedImmune and the investigators).

Gastrointestinal abnormalities including:

refractory nausea and vomiting, inability to take oral medication; requirement for intravenous alimentation; prior surgical procedures affecting absorption including total gastric resection; treatment for active peptic ulcer disease in the past 6 months; active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 120 days without evidence of resolution documented by endoscopy or colonoscopy; malabsorption syndromes. Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors, or inducers or substrates for CYP1A2 (see Section 10.8, concomitant therapy).

Concomitant medications known to prolong the QT interval (see Appendices 4, 5 and 6, concomitant therapy) or with factors that increase the risk of QTc prolongation or risk of arrhythmic events (such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age), history of Torsades de pointes.

Poorly controlled hypertension (persistently elevated > 150/100mmHg, either systolic or diastolic or both, despite anti-hypertensive medication) ECG with mean resting QTc of ≥470ms (Fridericia; as per local reading) on two or more time points within a 24 hour period or family history of long QT syndrome.

Requirement of anticoagulant therapy with oral vitamin K antagonists. Therapeutic use of low molecular weight heparin is allowed.

Any of the following within 12 months prior to study entry:

myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, Peripheral arterial embolus.

Active or prior documented autoimmune or inflammatory disorders (except vitiligo), for example:

Intestinal: Inflammatory Bowel Disease (Colitis (including ulcerative colitis), Crohn's Disease), Diverticulitis (with the exception of Diverticulosis), Coeliac Disease (except patients with coeliac disease controlled by diet alone), irritable Bowel Disease Vascular: any type of vasculitic disorder, e.g. Wegener syndrome, granulomatosis with polyangiitis.

Endocrine: any endocrine alteration related to an autoimmune process e.g. Hashimoto syndrome, Grave's disease. NOTE: patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement treatment may be included.

Respiratory: Active Pneumonitis (of any origin: inflammatory or infectious), Sarcoidosis syndrome.

Dermatological: Psoriasis, Lupus/SLE (unless the skin condition has never required systemic therapy).

Other: Rheumatoid Arthritis, Hypophysitis, Uveitis. History of organ transplant that requires use of immunosuppressive medications or any medical condition in which immunosuppressive agents were administered, including but, not limited to: Systemic corticosteroids, methotrexate, azathioprine.

Tumour necrosis factor alpha (TNF-α) blockers Patients with autoimmune conditions without active disease in the past 5 years may be included but only after discussion with the Study Physician.

Current or prior use of immunosuppressive agents within 28 days of first day of study drug, with the exceptions of intranasal or inhaled corticosteroids, or systemic corticosteroids at physiological doses which are not to exceed 10mg/day prednisolone (or an equivalent corticosteroid). The following exceptions are allowed:

Intranasal, inhaled, topical or local steroid injections (e.g. intra articular injection).

Systemic corticosteroids at physiological doses not to exceed 10mg/day prednisolone (or equivalent).

Steroids for premedication of hypersensitivity reactions (e.g. as CT premedication) .

Immunocompromised patients (e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV), or have a history of active primary immunodeficiency).

Previous allogeneic bone marrow transplant or double umbilical cord blood transplantation.

Receipt of live, attenuated vaccine within the last 30 days. Note: enrolled patients should not receive live vaccine while receiving investigational agent nor within 30 days of last dose of investigational agent.

Active infection including tuberculosis (clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV1/2 antibodies).

Subjects with a past or resolved HBV infection (defined as: presence of hepatitis B core antibody -anti-HBc- and absence of hepatitis B surface antigen -HbsAg-) are eligible.

As judged by the Investigator, any patient considered a poor medical risk due to a serious uncontrolled medical or psychiatric disorder, non-malignant systemic disease or on-going or active infection.

Persistent toxicities (≥Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia and vitiligo.

Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.

For Durvalumab-containing arms only: Patient with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the investigator.

Women who are pregnant, or are lactating or breastfeeding. Women of childbearing potential and male participants who are unwilling to use adequate contraception from screening and for 180 days after the last dose of study drug.

Patients with contraindication to MRI including; contraindicated metallic implants, contraindicated coronary stents and pacemakers. Inability to lie flat or still in an MRI scanner for whatever reason (e.g. claustrophobia) Judgement by the Investigator that the patient should not participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Proof-of-Mechanism (ktrans): to assess for 30% ktrans change between pre-IMP treatment and IMP End of Treatment DCE-MRI | Change between Screening and 72 hours before surgery
  Cediranib and Olaparib single IMP, Cediranib and Olaparib in combination IMP arms, having received at least 14 days' worth of IMP
Proof-of-Mechanism (CD8): to assess for 30% change between pre-IMP treatment and IMP End of Treatment in CD8 positive T-cells. This will be based on IHC assessment via histoscore | Change between Screening and 72 hours before surgery
  Durvalumab single IMP, durvalumab and olaparib combination IMP arms. having received at least 14 days' worth of IMP. Also assessed on D14 of IMP

SECONDARY OUTCOMES:
Number of participants with, and severity of, Adverse Events | From consent to 3 months post-surgery
  AEs are graded for severity according to the CTCAE toxicity criteria (Version 5.0)
Change in primary tumour size assessed by DCE-MRI | Between days -28 to 0 and 72 hrs before surgery, having received at least 2 weeks' worth of IMP
  Change in primary tumour size assessed by DCE-MRI
Tumour Response | Between days -28 to 0 for all patients.At 72 hrs before surgery if metastases are present,having received at least 2 wks' worth of IMP).Then every 8 wks until end of study (study ends=3 mths post surgery) or until progression
  Assessment of tumour response according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Grant D Stewart, Study Chair — Cambridge University Hospitals NHS Foundation Trust & University of Cambridge; Brent O'Carrigan, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust & University of Cambridge
Locations (2):
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge, England
  - Beatson Institute for Cancer Research, Glasgow

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Horvat-Menih I, McLean MA, Birchall J, Zamora Morales MJ, Wylot M, Ursprung S, Woitek R, Serrao E, Grimmer A, Latimer E, Khan AS, Priest AN, Gill AB, Kaggie JD, Graves MJ, Barrett T, Wason JM, Mossop H, Thomas M, Said S, Warren AY, Fife K, Eisen T, Matakidou A, Ince W, O'Carrigan B, Jones JO, Welsh SJ, Mitchell TJ, Armitage JN, Riddick AC, Stewart GD, Gallagher FA. Evaluating the metabolic effects of neoadjuvant treatment in clear cell renal cell carcinoma using hyperpolarized [1-13 C]pyruvate MRI. Abdom Radiol (NY). 2025 Dec 10. doi: 10.1007/s00261-025-05313-z. Online ahead of print. PMID 41369900
- [Derived] Horvat-Menih I, Li H, Priest AN, Li S, Gill AB, Mendichovszky IA, Francis ST, Warren AY, O'Carrigan B, Welsh SJ, Jones JO, Riddick ACP, Armitage JN, Mitchell TJ, Stewart GD, Gallagher FA. High-resolution and highly accelerated MRI T2 mapping as a tool to characterise renal tumour subtypes and grades. Eur Radiol Exp. 2024 Jul 10;8(1):76. doi: 10.1186/s41747-024-00476-8. PMID 38981998
- [Derived] Ursprung S, Mossop H, Gallagher FA, Sala E, Skells R, Sipple JAN, Mitchell TJ, Chhabra A, Fife K, Matakidou A, Young G, Walker A, Thomas MG, Ortuzar MC, Sullivan M, Protheroe A, Oades G, Venugopal B, Warren AY, Stone J, Eisen T, Wason J, Welsh SJ, Stewart GD. The WIRE study a phase II, multi-arm, multi-centre, non-randomised window-of-opportunity clinical trial platform using a Bayesian adaptive design for proof-of-mechanism of novel treatment strategies in operable renal cell cancer - a study protocol. BMC Cancer. 2021 Nov 18;21(1):1238. doi: 10.1186/s12885-021-08965-4. PMID 34794412